CLINICAL TRIAL: NCT06253962
Title: Carotid Atherosclerosis in Predicting Coronary Artery Disease
Acronym: CACA
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CACA
Record Dates: First submitted 2024-02-04; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Carotid Atherosclerosis; Coronary Atheroscleroses
MeSH Terms: conditions — Carotid Artery Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- carotid atherosclerosis
  Interventions: Other: coronary agiongraphy
- without carotid atherosclerosis
  Interventions: Other: coronary agiongraphy

INTERVENTIONS:
Other: coronary agiongraphy — severity of coronary atherosclerosis

SUMMARY:
Carotid plaque burden and composition features, particularly lipid necrotic core, are significantly associated with severity of CAD stenosis. This study aims to explore the relationship between various phenotypic patterns of carotid atherosclerosis with the prevalence, phenotype, and severity of coronary atherosclerosis. The patients with chest tightness or chest pain will receive carotid artery ultrasonography before coronary angiography so as to explore the relationship between them.

ELIGIBILITY:
Inclusion Criteria:

* patients receive carotid ultrasound and coronary angiography

Exclusion Criteria:

* None

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to receive coronary angiography. Carotid ultrasound performed before angiography.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | two years after angiography
  acute myocardial infarction; heart failure; cardiac death; revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided